CLINICAL TRIAL: NCT06407726
Title: Comparative Effects of Virtual Reality and Vestibular Exercises on Balance, Gait, and Activities of Daily Living in Older Adults
Brief Title: Comparative Effects of Virtual Reality and Vestibular Exercises on Balance Gait in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0280
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Old Age; Vestibular Disorder; Balance; Exercise
Keywords: Old Age; Vestibular Disorder; Balance; Exercise
MeSH Terms: conditions — Vestibular Diseases; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomized through lottery method and allocated into two groups. Group A (n=22) participants will receive Virtual Reality intervention with conventional treatment, while Group B (n=22) will receive Vestibular Exercises with conventional treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- participants will receive Virtual Reality intervention with conventional treatment, (Experimental): Participants will receive 40-minute sessions five days per week for six weeks of Virtual Reality intervention and conventional therapy.
  Interventions: Other: virtual reality training group
- participants will receive Vestibular Exercises with conventional treatment. (Active Comparator): Participants will receive 40-minute sessions five days per week for six weeks of Vestibular Exercises and conventional therapy.
  Interventions: Other: vestibular exercise group

INTERVENTIONS:
Other: virtual reality training group — Participants will receive 40-minute sessions five days per week for six weeks of Virtual Reality intervention and conventional therapy.
  Arms: participants will receive Virtual Reality intervention with conventional treatment,
Other: vestibular exercise group — Participants will receive 40-minute sessions five days per week for six weeks of Vestibular Exercises and conventional therapy.
  Arms: participants will receive Vestibular Exercises with conventional treatment.

SUMMARY:
To compare the effects of virtual reality and vestibular exercises on balance, gait, and activities of daily living in older adults.

DETAILED DESCRIPTION:
It will be a randomized clinical trial where non-probability convenience sampling technique will be used. Total 44 participants will be taken aged 60 to 85 years. All Participants will be randomized through lottery method and allocated into two groups. Group A (n=22) participants will receive Virtual Reality intervention with conventional treatment, while Group B (n=22) will receive Vestibular Exercises with conventional treatment. The Berg Balance Scale for balance assessment, Dynamic Gait Index for gait while Time Up and Go Test, and Modified Barthel Index for Activities of Daily Living will be outcome measure tools.

ELIGIBILITY:
Inclusion Criteria:

* Older adults with or without any assistive device.
* Participants with a Mini-Mental State Examination score greater than 24.
* Participants with a value greater than 10 secs on the Time Up and Go Test.

Exclusion Criteria:

* Severe visual or vestibular impairments (e.g., Meniere's disease, labyrinthitis).
* Significant musculoskeletal impairments (e.g., arthritis, joint contractures).
* Unstable medical conditions (e.g., uncontrolled hypertension, cardiovascular disease).
* History of epilepsy or seizures.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
The Dynamic Gait Index (DGI) | 6 months
  The Dynamic Gait Index (DGI) is a clinical tool assessing balance during walking under different external conditions. It uses a four-point ordinal scale, with a total score of 24. Scores below 19 indicate a higher risk of falls in older adults, while scores above 22 suggest safe ambulation. The DGI has demonstrated validity as a measure of functional mobility and strongly predicts falls
Berg Balance Scale | 6 months
  Berg Balance Scale: is a clinical tool assessing static and dynamic balance through 14 functional tasks, each scored from 0 to 4, with a maximum score of 56. Scores below 45 indicate a higher risk of falling. It has demonstrated excellent validity, correlating well with the Timed Up-and-Go test. It also exhibits excellent test-retest reliability, making it a widely accepted tool for measuring balance and mobility.
Modified Barthel Index | 6 months
  Modified Barthel Index is widely accepted measure of physical disability, assessing activities of daily living. Scoring ranges from 0 to 20, with lower scores indicating increased disability. The total score reflects the patient's independence in daily activities, with changes of more than two points indicating a probable genuine change. The index has demonstrated validity, with scores between 0.73 and 0.77 compared to a motor ability index for stroke patients.It also exhibits high inter-rater and test-retest reliability,Higher scores indicates maximum recovery

CONTACTS AND LOCATIONS:
Overall Officials: Zeest hashmi, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tornero-Quinones I, Saez-Padilla J, Espina Diaz A, Abad Robles MT, Sierra Robles A. Functional Ability, Frailty and Risk of Falls in the Elderly: Relations with Autonomy in Daily Living. Int J Environ Res Public Health. 2020 Feb 5;17(3):1006. doi: 10.3390/ijerph17031006. PMID 32033397
- [Background] Nobrega-Sousa P, Gobbi LTB, Orcioli-Silva D, Conceicao NRD, Beretta VS, Vitorio R. Prefrontal Cortex Activity During Walking: Effects of Aging and Associations With Gait and Executive Function. Neurorehabil Neural Repair. 2020 Oct;34(10):915-924. doi: 10.1177/1545968320953824. Epub 2020 Aug 31. PMID 32865134
- [Background] Lockie RG, Dawes JJ, Kornhauser CL, Holmes RJ. Cross-Sectional and Retrospective Cohort Analysis of the Effects of Age on Flexibility, Strength Endurance, Lower-Body Power, and Aerobic Fitness in Law Enforcement Officers. J Strength Cond Res. 2019 Feb;33(2):451-458. doi: 10.1519/JSC.0000000000001937. PMID 28445229